CLINICAL TRIAL: NCT07040280
Title: A Phase II Double-Blind Trial of Sulforaphane for Therapeutic Prevention of Melanoma in Patients With Multiple Atypical Nevi and a Prior History of Melanoma
Brief Title: Testing the Effect of Sulforaphane, a Compound Naturally Found in Cruciferous Vegetables, on Preventing Melanoma in Patients With a Prior History of Melanoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EA6232; HT94252311028 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2025-06-17; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Melanoma
Keywords: Melanoma; Skin Neoplasm
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — sulforaphane

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- A (Experimental): Three tablets of Avmacol® Extra Strength [Nutramax] by mouth, once daily, for 12 months
  Interventions: Drug: Sulforaphane (broccoli sprout extract); Device: Derma-AI
- B (Placebo Comparator): Placebo - Three tablets by mouth, once daily, for 12 months
  Interventions: Drug: Placebo; Device: Derma-AI

INTERVENTIONS:
Drug: Sulforaphane (broccoli sprout extract) — Sulforaphane - Three tablets of Avmacol® Extra Strength [Nutramax] by mouth, once daily, for 12 months.
  Other Names: (Avmacol® Extra Strength)
  Arms: A
Drug: Placebo — Three tablets by mouth, once daily, for 12 months
  Arms: B
Device: Derma-AI — Photographs of lesions as part of the clinical exam at baseline, three (3) months, and twelve (12) months. These photographs will be submitted for assessment by a software called Derma-AI, which tracks moles over time for changes in size, number, and appearance

SUMMARY:
The goal of this clinical trial is to compare the safety and effects of sulforaphane with the safety and effects of placebo on people's risk of developing melanoma. The main question it aims to answer is:

Will giving sulforaphane (a broccoli sprout extract) have a meaningful effect on how your atypical moles change over time? If there is an effect, will this lower your risk of developing melanoma?

Participants will:

Take sulforaphane or a placebo for 12 months Visit the clinic once every 3 months for checkups and tests You will keep a calendar which will help you keep track of when you take your tablets

ELIGIBILITY:
Inclusion Criteria:

* Patient must have ≥ 3 clinically atypical nevi, assessed within 30 days prior to randomization, that are consistent with the International Agency for Research on Cancer (IARC) definition as follows.27
* Must have a diameter of ≥ 5mm in one dimension
* Must include a macular component in at least one area
* Must have at least two of the following features: ill-defined borders, color variegation, uneven contour, and erythema
* Patient must have a prior diagnosis of early-stage melanoma, defined as either melanoma in situ, localized resected stage I-II node negative melanoma, or resected node positive stage III melanoma who in the assessment of their physician have a low risk of relapse of their prior melanoma within one year of randomization.
* Patient must not be currently on targeted or checkpoint immunotherapy or treated within 365 days prior to randomization.
* Patient must be ≥ 18 years of age.
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with a prior or concurrent malignancy (other than the melanoma for which they are on this study), whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen, are eligible for this trial.

Exclusion Criteria:

* Patient must not be pregnant.
* Patient must not have a known allergy to cruciferous vegetables.
* Patients must not use any other sulforaphane-containing dietary supplement during the study period.
* Patient must not be on any current systemic treatment for melanoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the total area of nevi after 12 months of treatment from the baseline between sulforaphane and placebo arms | 12 months of treatment
  The change in the total area of atypical and common pigmented nevocellular nevi measured at baseline and after 12 months of treatment, will be assessed in each patient who completed the full 12 months of treatment (with compliance assessed by dosing logs). The difference in the change of total area of nevi between the two arms will be compared using the Wilcoxon rank sum test.

SECONDARY OUTCOMES:
Change in number of atypical nevi at baseline and after the last treatment be assessed via automated image analysis | After 12 months of treatment
  The number of changed atypical nevi at baseline and after the last treatment (12 months) will be assessed via automated image analysis. The difference in baseline and post-treatment measures will be compared between the two arms using the Wilcoxon rank-sum test.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Over 12 months
  Toxicity rate for individual AEs, categorized AEs and worst degree AEs will be compared between the two arms using the Fisher's exact test

OTHER OUTCOMES:
Effects of Sulforaphane on Inflammation and Immunity | Baseline and 3 months and also baseline and 12 month
  Analysis of circulating cytokines, the Wilcoxon signed-rank test will be used to compare the level of each value between timepoints. The Wilcoxon rank-sum test will be used to compare changes in levels between patients receiving sulforaphane and placebo between baseline and 3 months and also baseline and 12 month timepoints.
Effects of Sulforaphane on Inflammation and Immunity | After 12 months
  Pre-post treatment comparisons of mRNA levels normalized to housekeeping genes will be performed using the Wilcoxon signed rank tests. Kruskal-Wallis test will be used to assess differential affects genes grouped into broad pathways as was previously described for sulforaphane
Effects of Sulforaphane on Inflammation and Immunity | After 12 months
  Dermoscopy and dermoscopic photographs will be performed on the index nevi at each timepoint, and morphologic features will be reported descriptively
Effects of Sulforaphane on Inflammation and Immunity | Baseline and 3 months and also baseline and 12 month
  Analysis of the semi-quantitative scoring of immune cell infiltration, the Wilcoxon signed-rank test will be used to compare the level of each value between timepoints. The Wilcoxon rank-sum test will be used to compare changes in levels between patients receiving sulforaphane and placebo between baseline and 3 months and also baseline and 12 month timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: John Kirkwood, MD, Study Chair — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States